CLINICAL TRIAL: NCT04591067
Title: Physical Capacity Among Patients Treated With Periacetabular Osteotomy for Hip Dysplasia: a Cross-sectional Study
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Sally Oppendieck Andersen, MSc. Human Physiology, BSc. Exercise & Sport Sciences, Copenhagen University Hospital, Hvidovre
Other Study IDs: 20006975
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Hip Dysplasia; Joint Diseases; Musculoskeletal Diseases
Keywords: Hip Dysplasia; Hip and muscle-tendon related groin pain; Musculoskeletal Diseases
MeSH Terms: conditions — Hip Dislocation; Joint Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hip Dysplasia group: Subjects who have undergone a periacetabular osteotomy (PAO) for hip dysplasia within the last 1-5 years.
  Interventions: Other: Testing of physical capacity

INTERVENTIONS:
Other: Testing of physical capacity — This cross-sectional study will involve evaluation of physical capacity by assessment of:
  1. Gait function
  2. Muscle activity during walking
  3. Endurance during walking
  4. Hip muscle strength
  5. Hip range of motion
  6. Hip and muscle-tendon-related groin pain
  7. Hip and groin related patient-reported outcome measures (PROMs)

SUMMARY:
This cross-sectional study investigates the physical capacity of patients, who have undergone a periacetabular osteotomy for hip dysplasia within the last 1-5 years.

DETAILED DESCRIPTION:
Hip dysplasia is a common disease both worldwide and among the Danish population. The disease is characterized by a shallow and oblique acetabulum, resulting in insufficient coverage of the femoral head. The abnormalities of the dysplastic hip joint lead to altered biomechanical adaptations, highly affecting the physical capacity of patients. Studies have shown that patients with hip dysplasia experience reduced muscle strength and gait abnormalities, when compared to healthy controls.

Each year, approximately 200 Danes with hip dysplasia are treated with periacetabular osteotomy (PAO). As the preferable joint-preserving surgical treatment for younger patients with symptomatic hip dysplasia, the PAO reduces prevalence of muscle-tendon-related pain and improves hip and groin related patient-reported outcome measures (PROMs). By extension, studies report a hip survival rate of approximately 75% 12 years following PAO.

However, little is known about objective measures of physical capacity following PAO. Despite reducing muscle-tendon-related pain and improving PROMs, gait adaptations still remain and studies report no improvements in muscle strength, nor in the physical activity profile, 1 year following treatment with PAO. Thus, the field calls for research aiming to identify parameters of impaired physical capacity in patients treated with PAO. Thorough knowledge of physical capacity in these patients may contribute to the establishment of a science-based rehabilitation strategy, potentially improving physical activity, function, work capacity and quality of life.

The primary aim of this study is to analyse and identify parameters of impaired physical capacity in patients with hip dysplasia 1-5 years following treatment with PAO. Gait function, defined as peak hip extension angle and peak hip flexor moment, is chosen as the primary outcome, due to previously shown correlations between the extent of gait impairments and the Copenhagen Hip and Groin Outcome Score (HAGOS).

As recommended by the International Hip-related Pain Research Network (IHiPRN), measurements of physical capacity in patients with hip-related pain should include: clinical measures, laboratory-based measures, measures of physical activity and return to physical activity. Secondary outcomes of this study are: muscle activity during level walking and walking with inclination, endurance and pain during walking, range of motion (ROM), muscle strength, hip and muscle-tendon-related pain, radiographic measures and PROMs (present level of physical activity and sports & activity level prior to and after treatment with PAO).

We hypothesise that patients with the lowest scores of HAGOS subscales pain and sport/recreation will have the lowest physical capacity, measured as: gait impairments, reduced muscle strength and prevalence of muscle-tendon-related pain.

This is a cross-sectional study.

Thirty subjects from across the country, aged 18-40 years, who have undergone a PAO for hip dysplasia within the last 1-5 years, will be included in the study.

All testing will be performed at Copenhagen University Hospital, Hvidovre.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40 years
* BMI < 30
* Primary diagnosis of ipsilateral or bilateral hip dysplasia
* Treated with PAO for hip dysplasia unilaterally or bilaterally within 1-5 years

Exclusion Criteria:

* Retroverted acetabulum (positive posterior wall sign and ischial spine sign) treated with reversed PAO
* Total Hip Arthroplasty (THA)
* Pain management with analgesics or other medication affecting muscle function and perception of pain
* A need for walking aids to be able to walk freely

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects who have undergone a periacetabular osteotomy (PAO) for hip dysplasia within the last 1-5 years.
  Subjects will be recruited through social media from two specific closed-member facebook groups for patients with hip dysplasia. Permission for recruiting through social media was granted by The Danish Data Protection Agency along with permission for the handling of personal data (P-2020-261).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Gait function | Baseline
  Peak hip extension angle and peak hip flexor moment

SECONDARY OUTCOMES:
Gait function following fatigue | Baseline
  Peak hip extension angle and peak hip flexor moment following a 6-Minute walk test
Muscle activity | Baseline
  Muscle activity of hip specific muscles during level walking and walking with inclination
Maximal voluntary isometric hip muscle force | Baseline
  Adduction, abduction, flexion and extension
Hip and muscle-tendon-related groin pain | Baseline
  FADIR and FABER, modified standardized clinical entity approach
Hip specific patient reported outcome measures (PROMs) | Baseline
  Present level of physical activity and sports & activity level prior to and after treatment with PAO

CONTACTS AND LOCATIONS:
Overall Officials: Per Hölmich, Professor, dr.med., Study Director — Sports Orthopedic Research Center - Copenhagen (SORC-C), Copenhagen University Hospital Amager-Hvidovre, Hvidovre, Denmark
Locations (1):
- Department of Orthopedic Surgery, Copenhagen University Hospital Amager-Hvidovre, Hvidovre, Denmark, Copenhagen, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Andersen SO, Ishoi L, Karabanov AN, Bencke J, Holmich P. Physical function in patients treated for hip dysplasia with periacetabular osteotomy and in some cases with supplementary hip arthroscopy: A cross-sectional study. Clin Biomech (Bristol). 2025 Dec;130:106677. doi: 10.1016/j.clinbiomech.2025.106677. Epub 2025 Oct 9. PMID 41138707